CLINICAL TRIAL: NCT04989192
Title: On Dose Efficiency of Modern CT-Scanners in the Staging of Malignancies - a Prospective Randomized Study
Brief Title: Dose Efficiency of Modern CT Scanners in Oncologic Scans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-0280
Record Dates: First submitted 2021-07-23; First posted 2021-08-04 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms; Neoplasm Metastasis; Metastatic Cancer
Keywords: Spectral CT; CT; Computed Tomography; Radiation Dose; Dose Efficiency
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Randomization of patients referred for a staging CT scan one of three CT scanners routinely used for this purpose in our department
Masking Description: no masking required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT scanner 1 (Other): Patients will undergo imaging on scanner 1.
  Interventions: Diagnostic Test: Scan at CT scanner 1
- CT scanner 2 (Other): Patients will undergo imaging on scanner 2.
  Interventions: Diagnostic Test: Scan at CT scanner 2
- CT scanner 3 (Other): Patients will undergo imaging on scanner 3.
  Interventions: Diagnostic Test: Scan at CT scanner 3

INTERVENTIONS:
Diagnostic Test: Scan at CT scanner 1 — Patients will undergo imaging on a modern CT scanner with spectral imaging capabilities. A dose neutral spectral acquisition mode will routinely be used. Contrast material protocol and scan ranges are similar among all three arms.
  Arms: CT scanner 1
Diagnostic Test: Scan at CT scanner 2 — Patients will undergo imaging on a modern 128 slice CT-scanner without spectral imaging capabilities. A standard acquisition protocol will be used. Contrast material protocol and scan ranges are similar among all three arms.
  Arms: CT scanner 2
Diagnostic Test: Scan at CT scanner 3 — Patients will undergo imaging on a modern 20 slice CT-scanner without spectral imaging capabilities. A standard acquisition protocol will be used. Contrast material protocol and scan ranges are similar among all three arms.
  Arms: CT scanner 3

SUMMARY:
CT-Staging is crucial for therapy planning of patients with malignancies. Dose efficiency and image quality are important parameters for these examinations. Up to now, scientific evidence of dose efficiency of modern CT scanners is mostly derived from retrospective analyses. This prospective study systematically analyzes dose efficiency and image quality of three modern CT scanners by randomization of patients who are scheduled for a CT scan to examine the status of malignancies. After giving informed consent and randomization (1:1:1), the CT scan will be performed at one of the modern CT scanners available at our department. This will allow a systematic allocation to the different scanners.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of a malignancy or known / confirmed malignancy AND
* indication for contrast-enhanced CT of the body confirmed by board-certified radiologist ('justifying indication' according to German/European radiation protection law) AND
* patient (is able to give informed consent and) has given informed consent.

Exclusion Criteria:

* age < 18 years
* known or suspected pregnancy
* contraindications for contrast agent (renal failure, allergy, hyperthyroidism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-08-17 (Estimated); Study Completion 2023-08-17 (Estimated)

PRIMARY OUTCOMES:
Objective Image Quality | 1 year
  measured as signal, noise and modulation transfer function equivalent parameters derived from patient scans
Radiation Dose | 1 year
  measured as x-ray tube parameters such as dose length product (DLP)

SECONDARY OUTCOMES:
Subjective Image Quality (entire cohort and for individual disease groups) | 1 year
  measured by blinded evaluation by radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Florian Schwarz, MD, Principal Investigator — Universitätsklinikum Augsburg
Locations (1):
- University Hospital Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data upon request (pending final approval by the data protection officer).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for sharing individual participant data will be considered at the time of publication of the first manuscript containing result data.
Access Criteria: We plan to share data on request at this point in time.

REFERENCES:
- [Derived] Risch F, Decker JA, Popp D, Sinzinger A, Braun F, Bette S, Jehs B, Haerting M, Wollny C, Scheurig-Muenkler C, Kroencke TJ, Schwarz F. Artifact Reduction From Dental Material in Photon-Counting Detector Computed Tomography Data Sets Based on High-keV Monoenergetic Imaging and Iterative Metal Artifact Reduction Reconstructions-Can We Combine the Best of Two Worlds? Invest Radiol. 2023 Sep 1;58(9):691-696. doi: 10.1097/RLI.0000000000000967. PMID 36897803